CLINICAL TRIAL: NCT04776616
Title: Green Light Therapy As a Non-Pharmacologic Intervention to Decrease Anxiety in Pregnant Women With Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011231501
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2021-02

CONDITIONS: Anxiety
Keywords: Pregnancy; Opioid Use Disorder; ACE; STAI
MeSH Terms: conditions — Anxiety Disorders; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized controlled trial with 1:1 control and intervention
Who Masked: Participant
Masking Description: Participants will choose a piece of folded paper from a container. This piece of paper will indicate whether they are receiving the control or the experimental intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to white LED light (Sham Comparator): Participants will be exposed to white LED strip lights in a dark room for 2 hours a day
  Interventions: Device: Exposure to white LED light
- Exposure to green LED light (Experimental): Participants will be exposed to green LED strip lights in a dark room for 2 hours a day.
  Interventions: Device: Exposure to green LED light

INTERVENTIONS:
Device: Exposure to white LED light — Participants will be exposed to white LED strip lights in a dark room for 2 hours a day
  Arms: Exposure to white LED light
Device: Exposure to green LED light — Participants will be exposed to green LED strip lights in a dark room for 2 hours a day
  Arms: Exposure to green LED light

SUMMARY:
This is a clinical trial evaluating anxiety reduction for women with opioid use disorder affecting pregnancy. It is well documented that anxiety increases as pregnancy progresses. The investigators hypothesize that women who undergo green light therapy (experimental arm) will have a smaller increase in anxiety scores compared to the women who undergo white light therapy (control arm).

The investigators will also look at how much opiate replacement therapy increases women require during the study period, and how much opiate they require during admission for delivery. The investigators think this a is a low risk intervention in a pregnant population that has higher levels of anxiety when compared to the general population. The investigators believe based on animal studies that this could be effective, and change the way providers treat and support individuals with substance use disorder.

The opioid epidemic has negatively impacted our society at many levels. Finding non-pharmacologic ways to support patients while in recovery/sustained sobriety that are simple and low cost would be a step forward in providing compassionate and comprehensive treatment to individuals affected by Opioid Use Disorder.

DETAILED DESCRIPTION:
At time of enrollment, participants will be administered a States-Traits Anxiety Inventory (STAI) questionnaire, undergo screening for ACE score (adverse childhood experiences), and will be asked about basic demographic data. After they complete the initial surveys, the patient will be assigned to either the control group or the experimental group. They will be sent home with the light, along with instructions to use their light every night for 1-2 hours as ambient lighting. The investigators hope to enroll a maximum of 26 patients in this study with 1:1 randomization (13 control, 13 experiment).

At approximately halfway through the intervention, the PI will call the patient and ask how often she has been using the light, how long she uses the light for every night, and whether she has noticed any effects (either positive or negative).

At the prenatal visit around 36 weeks gestation or at time of delivery, whichever is sooner, patients will be asked by the PI to turn in their light and also fill out the STAI once again.

After delivery, the PI will review the medical record and record any change in opioid replacement therapy during pregnancy as well as the total dose of opiate required during the inpatient admission for delivery.

The investigators hope to enroll a maximum of 26 patients in this study with 1:1 randomization (13 control, 13 experiment)

ELIGIBILITY:
Inclusion Criteria:

Pregnant women between 20 - 32 weeks gestation with a diagnosis of opiate use disorder receiving care through Banner University Medical Center North Mothers Over Medicine (MOMs) Clinic, a high-risk pregnancy clinic for women with substance use disorder complicating pregnancy

Exclusion Criteria:

1. Inability to speak or understand English
2. Incarcerated individuals
3. Age <18 yo

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in anxiety over course of intervention, measured by STAI | 4-16 weeks
  The participants will be given a States-Traits Anxiety Inventory (STAI) questionnaire at time of enrollment and then again at time of completion. Score range is 20 to 80, with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Change in Opiate Replacement Therapy | 4-20 weeks
  The participants dose of opiate replacement therapy will be recorded at time of enrollment, at time of completion of the study, and also at time of delivery if it doesn't coincide with completion of study.
Opiate used during admission for delivery | 1-7 days
  The participants total dose of opiate administered during the admission for delivery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Miller, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner North Clinic, Obstetrics & Gynecology Clinic, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibrahim MM, Patwardhan A, Gilbraith KB, Moutal A, Yang X, Chew LA, Largent-Milnes T, Malan TP, Vanderah TW, Porreca F, Khanna R. Long-lasting antinociceptive effects of green light in acute and chronic pain in rats. Pain. 2017 Feb;158(2):347-360. doi: 10.1097/j.pain.0000000000000767. PMID 28092651
- [Background] Gros DF, Milanak ME, Brady KT, Back SE. Frequency and severity of comorbid mood and anxiety disorders in prescription opioid dependence. Am J Addict. 2013 May-Jun;22(3):261-5. doi: 10.1111/j.1521-0391.2012.12008.x. PMID 23617869
- [Background] Ecker J, Abuhamad A, Hill W, Bailit J, Bateman BT, Berghella V, Blake-Lamb T, Guille C, Landau R, Minkoff H, Prabhu M, Rosenthal E, Terplan M, Wright TE, Yonkers KA. Substance use disorders in pregnancy: clinical, ethical, and research imperatives of the opioid epidemic: a report of a joint workshop of the Society for Maternal-Fetal Medicine, American College of Obstetricians and Gynecologists, and American Society of Addiction Medicine. Am J Obstet Gynecol. 2019 Jul;221(1):B5-B28. doi: 10.1016/j.ajog.2019.03.022. Epub 2019 Mar 27. No abstract available. PMID 30928567
- [Background] Newham JJ, Westwood M, Aplin JD, Wittkowski A. State-trait anxiety inventory (STAI) scores during pregnancy following intervention with complementary therapies. J Affect Disord. 2012 Dec 15;142(1-3):22-30. doi: 10.1016/j.jad.2012.04.027. Epub 2012 Sep 7. PMID 22959685
- [Background] Dube SR, Felitti VJ, Dong M, Chapman DP, Giles WH, Anda RF. Childhood abuse, neglect, and household dysfunction and the risk of illicit drug use: the adverse childhood experiences study. Pediatrics. 2003 Mar;111(3):564-72. doi: 10.1542/peds.111.3.564. PMID 12612237
- [Background] Anda RF, Brown DW, Felitti VJ, Dube SR, Giles WH. Adverse childhood experiences and prescription drug use in a cohort study of adult HMO patients. BMC Public Health. 2008 Jun 4;8:198. doi: 10.1186/1471-2458-8-198. PMID 18533034
- [Background] Stein MD, Conti MT, Kenney S, Anderson BJ, Flori JN, Risi MM, Bailey GL. Adverse childhood experience effects on opioid use initiation, injection drug use, and overdose among persons with opioid use disorder. Drug Alcohol Depend. 2017 Oct 1;179:325-329. doi: 10.1016/j.drugalcdep.2017.07.007. Epub 2017 Aug 5. PMID 28841495

DOCUMENTS (1):
  • Informed Consent Form (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT04776616/ICF_000.pdf